CLINICAL TRIAL: NCT01946516
Title: A Sero-Epidemiologic Survey and Cost Effectiveness Study of Screening for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) Among Newly Diagnosed Cancer Patients
Brief Title: S1204, Viral Screening in Newly Diagnosed Cancer Patients
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S1204; NCI-2013-01631 (Other: NCI); U10CA032102 (NIH)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: viral screening
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen submission is optional.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to estimate the prevalence of HIV, Hepatitis B and hepatitis C infection among newly diagnosed cancer patients presenting to community and academic oncology clinics.

DETAILED DESCRIPTION:
Primary Objective

Among newly diagnosed cancer patients presenting to SWOG-affiliated community and academic oncology clinics, estimate the prevalence of human immunodeficiency virus (HIV), hepatitis B (HBV), and hepatitis C (HCV) infection. Prevalence estimates will be further stratified: by whether infection with the virus(es) is known, as reported by patients and/or their physician prior to study testing, vs. unknown; by presenting cancer type, and by self-reported risk factors for each virus.

Secondary Objectives

* Evaluate known sociodemographic, clinical, and behavioral factors that are significantly associated with previously undiagnosed HIV, HBV, and/or HCV infection in a population of people with newly diagnosed cancer.
* Among patients who are identified as having HIV, HBV, and/or HCV, evaluate the timing and type of treatments received, both for the viral infections and the cancers.
* Evaluate type and rate of cancer treatment-related adverse events in patients with HIV, HBV, and/or HCV infection.
* Using simulation modeling that is directly informed by the data obtained from this study, determine the cost-effectiveness (expressed as cost per infection detected and cost per year of life gained) of (1) routine, universal screening and (2) risk factor-directed screening of newly diagnosed cancer patients for HIV, HBV, and/or HCV vs. current care.

Tertiary Objective

Create a biorepository of stored serum for future translational medicine studies that may include identifying genomic and viral factors that increase the risk of serious adverse effects among participants infected with HIV, HBV, and/or HCV being treated for invasive cancers.

ELIGIBILITY:
Inclusion Criteria:

* presenting for evaluation or treatment of a new cancer malignancy(including hematologic)
* confirmed pathologic diagnosis must be within 120 days of registration (Patients presenting for "second opinions" of confirmed malignancies are eligible, including those who have started cancer treatment at other facilities)
* at least 18 years of age
* patient must have had their blood drawn for HIV, HBV and HCV testing prior to registration (Patients who have had HIV, HBV and/or HCV testing within 60 days prior to registration and who do not wish to be retested are eligible, provided supporting documents can be obtained confirming viral test results for all three viruses. Documentation must be obtained prior to registration.

Patients who are viral positive for either HIV, HBV, and/or HCV and who do not wish to be retested are eligible, provided documentation of viral load within 120 days prior to registration can be obtained. Note that these patients must be tested for or provide current viral load for all three viruses to be eligible. Documentation must be obtained prior to registration.)

* Patients must sign and give written informed consent in accordance with institutional and federal guidelines
* Patients must be offered the opportunity to allow their blood specimens to be banked by the SWOG Repository for future research

Exclusion Criteria:

* diagnosed with a malignancy other than the current malignancy within the past five years (with the exception of basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ breast cancer.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community and academic oncology clinics
Sampling Method: Non-Probability Sample
Enrollment: 3051 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Ramsey, M.D., Study Chair — Fred Hutchinson Cancer Center
Locations (58):
- United States (58):
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Contra Costa Regional Medical Center, Martinez, California
  - East Bay Physicians Medical Group-Summit, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Mac Neal Hospital, Berwyn, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Veteran Administration Eastern Kansas Healthcare, Leavenworth, Kansas
  - Topeka VA Hospital, Topeka, Kansas
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - North Shore Hematology Oncology Associates Inc, Slidell, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - OneHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3092 participants were screened for the trial; 41 were deemed ineligible and 3051 eligible participants were registered to the trial.
Groups:
- HBV, HCV, or HIV Prevalence: Participants received testing for at least one of the following, HBV, HCV, or HIV.
Period: Overall Study
Arm/Group | HBV, HCV, or HIV Prevalence
Started | 3051
Evaluated for HBV Status | 3050
Evaluated for HCV Status | 2990
Evaluated for HIV Status | 3045
Completed | 3051
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes the 3051 participants that were eligible to receive at least one viral test.
Groups:
- Participants With Newly Diagnosed Cancer: Participants with newly diagnosed cancer that underwent viral testing for at least one of the following: HBV, HCV, and HIV.
Arm/Group | Participants With Newly Diagnosed Cancer
Number analyzed (Participants) | 3051
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1967
  >=65 years | 1084
Age, Continuous [Median (Full Range); unit: years] | 60.6 [18.2 to 93.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1842
  Male | 1209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 558
  Not Hispanic or Latino | 2478
  Unknown or Not Reported | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2281
  Race: Black | 553
  Race: Asian | 102
  Race: Other | 115
Cancer Type [Count of Participants; unit: Participants]
  Blood or marrow | 369
  Breast | 1058
  Gastrointestinal tract, colorectal | 362
  Gastrointestinal, liver | 62
  Gastrointestinal, other | 235
  Head and neck | 112
  Lung | 356
  Prostate | 100
  Other | 392
  Missing | 5
Region [Count of Participants; unit: Participants]
  West and Midwest United States | 1096
  South and Northeast United States | 1955

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Viral Infection
Description: An estimate of the prevalence of human immunodeficiency virus (HIV), hepatitis B (HBV), and hepatitis C (HCV) infection among newly diagnosed cancer participants presenting to SWOG-affiliated community and academic oncology clinics.
Time Frame: Up to 21 days after registration
Population: The analysis population includes the 3051 participants eligible to receive at least one viral test (for HBV, HCV, or HIV). 3050 participants were evaluable for HBV analysis (1 participants had no HBV test results available), 2990 participants were evaluable for HCV analysis (5 participants had no HCV test results available and 56 participants incomplete test results), and 3045 participants were evaluable for HIV analysis (6 participants had no HIV test results available).
Measure: Count of Participants; unit: Participants
Groups:
- Evaluated for Chronic HBV: Participants who were evaluated for chronic HBV.
- Evaluated for Previous HBV: Participants who were evaluated for previous HBV analysis.
- Evaluated for HCV: Participants who were evaluated for HCV..
- Evaluated for HIV: Participants who were evaluated for HIV analysis.
Arm/Group | Evaluated for Chronic HBV | Evaluated for Previous HBV | Evaluated for HCV | Evaluated for HIV
Number analyzed (Participants) | 3050 | 3050 | 2990 | 3045
Participants
  Positive Viral Test in All Participants | 19 | 197 | 71 | 34
  Positive Viral Test in Previously Diagnosed Participants | 11 | 25 | 49 | 32
  Positive Viral Test in Newly Diagnosed Participants | 8 | 172 | 22 | 2
  Positive Viral Test in Participants with Blood/Marrow Cancer: number analyzed (Participants) | 369 | 369 | 364 | 369
  Positive Viral Test in Participants with Blood/Marrow Cancer | 2 | 16 | 9 | 7
  Positive Viral Test in Participants with Breast Cancer: number analyzed (Participants) | 1058 | 1058 | 1046 | 1056
  Positive Viral Test in Participants with Breast Cancer | 4 | 66 | 9 | 2
  Positive Viral Test in Participants with Colorectal Cancer: number analyzed (Participants) | 362 | 362 | 356 | 362
  Positive Viral Test in Participants with Colorectal Cancer | 2 | 18 | 7 | 5
  Positive Viral Test in Participants with Liver Cancer: number analyzed (Participants) | 62 | 62 | 52 | 61
  Positive Viral Test in Participants with Liver Cancer | 4 | 5 | 9 | 0
  Positive Viral Test in Participants with GI, Other Tract Cancer: number analyzed (Participants) | 235 | 235 | 228 | 235
  Positive Viral Test in Participants with GI, Other Tract Cancer | 3 | 22 | 3 | 5
  Positive Viral Test in Participants with Head and Neck Cancer: number analyzed (Participants) | 111 | 111 | 106 | 111
  Positive Viral Test in Participants with Head and Neck Cancer | 1 | 9 | 5 | 1
  Positive Viral Test in Participants with Lung Cancer: number analyzed (Participants) | 356 | 356 | 347 | 356
  Positive Viral Test in Participants with Lung Cancer | 2 | 31 | 17 | 4
  Positive Viral Test in Participants with Prostate Cancer: number analyzed (Participants) | 100 | 100 | 98 | 100
  Positive Viral Test in Participants with Prostate Cancer | 0 | 12 | 3 | 1
  Positive Viral Test in Participants with Other Cancer: number analyzed (Participants) | 392 | 392 | 388 | 390
  Positive Viral Test in Participants with Other Cancer | 1 | 18 | 9 | 9

2. Secondary Outcome: Presence of Important Risk Factors in Participants Tested for Previous HBV
Description: The presence or absence of specific risk factors among participants evaluated for previous HBV is evaluated.
Time Frame: Up to 21 days after registration
Population: The analysis population includes the 2940 of the 3050 participants who were evaluable for HBV analysis and completed the risk factor survey.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Previous HBV Positive: Participants with previous HBV diagnosis.
- Participants With Previous HBV Negative: Participants without previous HBV diagnosis.
Arm/Group | Participants With Previous HBV Positive | Participants With Previous HBV Negative
Number analyzed (Participants) | 190 | 2750
Participants
  Sexual contact with HIV-positive person: Risk Factor Present | 14 | 25
  Sexual contact with HIV-positive person: Risk Factor Absent | 176 | 2725
  Self-reported infection with HCV or HIV: Risk Factor Present | 41 | 135
  Self-reported infection with HCV or HIV: Risk Factor Absent | 149 | 2615
  Born in high HBV prevalence region: Risk Factor Present | 63 | 243
  Born in high HBV prevalence region: Risk Factor Absent | 127 | 2507
  Injected drug use: Risk Factor Present | 21 | 86
  Injected drug use: Risk Factor Absent | 169 | 2664
  Unprotected sex with high-risk person: Risk Factor Present | 21 | 109
  Unprotected sex with high-risk person: Risk Factor Absent | 169 | 2641
  Sexual contact with hepatitis-positive person: Risk Factor Present | 10 | 56
  Sexual contact with hepatitis-positive person: Risk Factor Absent | 180 | 2694
  Unprotected sex with MSM, multiple, or anonymous partners: Risk Factor Present | 14 | 103
  Unprotected sex with MSM, multiple, or anonymous partners: Risk Factor Absent | 176 | 2647
  Diagnosis or treatment for STD: Risk Factor Present | 32 | 276
  Diagnosis or treatment for STD: Risk Factor Absent | 158 | 2474
  Blood transfusion between 1978-1985: Risk Factor Present | 13 | 110
  Blood transfusion between 1978-1985: Risk Factor Absent | 177 | 2640
  Needle-stick exposure: Risk Factor Present | 12 | 136
  Needle-stick exposure: Risk Factor Absent | 178 | 2614
  Household contact with hepatitis-positive person: Risk Factor Present | 15 | 171
  Household contact with hepatitis-positive person: Risk Factor Absent | 175 | 2579
  High-risk occupation: Risk Factor Present | 11 | 190
  High-risk occupation: Risk Factor Absent | 179 | 2560
  Completed HBV vaccine (3 or more doses): Risk Factor Present | 8 | 236
  Completed HBV vaccine (3 or more doses): Risk Factor Absent | 182 | 2514

3. Secondary Outcome: Presence of Important Risk Factors in Participants Tested for Chronic HBV
Description: The presence or absence of specific risk factors among participants evaluated for chronic HBV is evaluated.
Time Frame: Up to 21 days after registration
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Chronic HBV Positive: Participants with Chronic HBV diagnosis.
- Participants With Chronic HBV Negative: Participants without Chronic HBV diagnosis.
Arm/Group | Participants With Chronic HBV Positive | Participants With Chronic HBV Negative
Number analyzed (Participants) | 18 | 2922
Participants
  Born in high HBV prevalence region: Risk Factor Present | 8 | 298
  Born in high HBV prevalence region: Risk Factor Absent | 10 | 2624
  Needle-stick exposure: Risk Factor Present | 3 | 145
  Needle-stick exposure: Risk Factor Absent | 15 | 2777
  Unprotected sex with MSM, multiple, or anonymous partners: Risk Factor Present | 2 | 115
  Unprotected sex with MSM, multiple, or anonymous partners: Risk Factor Absent | 16 | 2807
  Unprotected sex with high-risk person: Risk Factor Present | 2 | 128
  Unprotected sex with high-risk person: Risk Factor Absent | 16 | 2794
  Sexual contact with hepatitis-positive person: Risk Factor Present | 1 | 65
  Sexual contact with hepatitis-positive person: Risk Factor Absent | 17 | 2857
  Diagnosis or treatment for STD: Risk Factor Present | 4 | 304
  Diagnosis or treatment for STD: Risk Factor Absent | 14 | 2618
  Self-reported infection with HCV or HIV: Risk Factor Present | 2 | 174
  Self-reported infection with HCV or HIV: Risk Factor Absent | 16 | 2748
  Household contact with hepatitis-positive person: Risk Factor Present | 1 | 185
  Household contact with hepatitis-positive person: Risk Factor Absent | 17 | 2737

4. Secondary Outcome: Presence of Important Risk Factors in Participants Tested for HCV
Description: The presence or absence of specific risk factors among participants evaluated for HCV is evaluated.
Time Frame: Up to 21 days after registration
Population: The analysis population includes the 2882 of the 2990 participants who were evaluable for HCV analysis completed the risk factor survey.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With HCV Positive: Participants with HCV diagnosis.
- Participants With HCV Negative: Participants without HCV diagnosis.
Arm/Group | Participants With HCV Positive | Participants With HCV Negative
Number analyzed (Participants) | 69 | 2813
Participants
  Injected drug use: Risk Factor Present | 21 | 67
  Injected drug use: Risk Factor Absent | 48 | 2746
  Tested because of blood exposure, injected drug use, or transfusion before 1992: Risk Factor Present | 9 | 45
  Tested because of blood exposure, injected drug use, or transfusion before 1992: Risk Factor Absent | 60 | 2768
  Tested because of symptoms: Risk Factor Present | 7 | 46
  Tested because of symptoms: Risk Factor Absent | 62 | 2767
  Blood transfusion between 1978-1985: Risk Factor Present | 11 | 104
  Blood transfusion between 1978-1985: Risk Factor Absent | 58 | 2709
  Tested because born between 1945-1965: Risk Factor Present | 11 | 126
  Tested because born between 1945-1965: Risk Factor Absent | 58 | 2687
  Self-reported infection with HIV: Risk Factor Present | 4 | 48
  Self-reported infection with HIV: Risk Factor Absent | 65 | 2765
  Snorted cocaine: Risk Factor Present | 15 | 254
  Snorted cocaine: Risk Factor Absent | 54 | 2559
  Needle-stick exposure: Risk Factor Present | 7 | 134
  Needle-stick exposure: Risk Factor Absent | 62 | 2679
  High-risk occupation: Risk Factor Present | 3 | 195
  High-risk occupation: Risk Factor Absent | 66 | 2618

5. Secondary Outcome: Presence of Important Risk Factors in Participants Tested for HIV
Description: The presence or absence of specific risk factors among participants evaluated for HIV is evaluated.
Time Frame: Up to 21 days after registration
Population: The analysis population includes the 2934 of the 3045 participants were evaluable for HIV analysis and completed the risk factor survey.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With HIV Positive: Participants with HIV diagnosis.
- Participants With HIV Negative: Participants without HIV diagnosis.
Arm/Group | Participants With HIV Positive | Participants With HIV Negative
Number analyzed (Participants) | 34 | 2900
Participants
  Sexual contact with HIV-positive person: Risk Factor Present | 16 | 23
  Sexual contact with HIV-positive person: Risk Factor Absent | 18 | 2877
  Unprotected sex with MSM, multiple, or anonymous partners: Risk Factor Present | 16 | 101
  Unprotected sex with MSM, multiple, or anonymous partners: Risk Factor Absent | 18 | 2799
  Diagnosis or treatment for STD: Risk Factor Present | 20 | 288
  Diagnosis or treatment for STD: Risk Factor Absent | 14 | 2612
  Unprotected sex with high-risk person: Risk Factor Present | 12 | 118
  Unprotected sex with high-risk person: Risk Factor Absent | 22 | 2782
  Self-reported infection with HBV: Risk Factor Present | 4 | 51
  Self-reported infection with HBV: Risk Factor Absent | 30 | 2849
  Diagnosis or treatment for tuberculosis: Risk Factor Present | 5 | 92
  Diagnosis or treatment for tuberculosis: Risk Factor Absent | 29 | 2808
  Injected drug use: Risk Factor Present | 3 | 104
  Injected drug use: Risk Factor Absent | 31 | 2796
  Needle-stick exposure: Risk Factor Present | 1 | 147
  Needle-stick exposure: Risk Factor Absent | 33 | 2753
  High-risk occupation: Risk Factor Present | 1 | 199
  High-risk occupation: Risk Factor Absent | 33 | 2701

6. Secondary Outcome: Type of Treatment for Cancer and Virus in Participants With Positive Viral Test
Description: Among participants with HIV, HBV, or HCV, the timing and type of treatments received, both for the viral infections and the cancers that were evaluated.
Time Frame: 60 days after registration
Population: The analysis population includes the 224 participants who were viral positive for at least one viral test (for HBV, HCV, or HIV) and had treatment outcome data available. Of the 292 patients were who were viral positive for at least one viral test, 11 patients did not have data submitted and 57 patients did not have data available.
Measure: Number; unit: percentage of participants
Groups:
- Participants With Previous HBV Infection: Participants with previous HBV diagnosis.
- Participants With Chronic HBV Infection: Participants with chronic HBV diagnosis.
- Participants With HCV Infection: Participants with previous HCV diagnosis.
- Participants With HIV Infection: Participants with previous HIV diagnosis.
- Participants With Any Type Of Viral Infection: Participants diagnosed with any type of viral infection.
Arm/Group | Participants With Previous HBV Infection | Participants With Chronic HBV Infection | Participants With HCV Infection | Participants With HIV Infection | Participants With Any Type Of Viral Infection
Number analyzed (Participants) | 152 | 15 | 49 | 30 | 224
percentage of participants
  Received Antiviral or Antiretroviral Drugs | 11.8 | 73.3 | 8.2 | 66.7 | 19.6
  Change in Cancer Treatment | 59.2 | 53.3 | 55.1 | 50 | 58.5
  Change in Cancer Treatment due to Viral Positive Status | 7.9 | 13.3 | 6.1 | 16.7 | 8
  Change in Cancer Treatment due to Viral Positive Status and Added Antiviral or Antiretroviral Drugs | 5.3 | 13.3 | 2 | 13.3 | 6.3

7. Secondary Outcome: Type and Rate of Adverse Events Among Patients With Viral Infection.
Description: Estimate type and rate of cancer-treatment related adverse events among persons with HIV, HBV, and/or HCV infection.
Time Frame: 5 years after registration
Reporting Status: Not Posted

8. Secondary Outcome: Cost-effectiveness of Viral Screening
Description: Estimate the cost-effectiveness of screening for HIV, HBV, and HCV.
Time Frame: 3 years after registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of study, 2 years.
Groups:
- HBV, HCV, or HIV Prevalence: Patients received testing for at least one of the following, HBV, HCV, or HIV,
Arm/Group | HBV, HCV, or HIV Prevalence
All-Cause Mortality (participants affected / at risk) | 0/3051
Serious Adverse Events (participants affected / at risk) | 0/3051
Other Adverse Events (participants affected / at risk) | 0/3051

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT01946516/Prot_SAP_ICF_000.pdf